CLINICAL TRIAL: NCT04692181
Title: Phase 1b/2a Evaluation of the Safety and Tolerability of SYN-004 in Adult Allogeneic Hematopoietic Cell Transplantation (Allo-HCT) Recipients
Brief Title: SYN-004 Safety and Tolerability in Allo-HCT Subjects
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theriva Biologics, Inc. (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: SB-1-004-006
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Acute Graft-Versus-Host Reaction Following Bone Marrow Transplant; Prevention of CDI in Adult Patients Being Treated With IV Beta-lactam Antibiotics
MeSH Terms: interventions — SYN-004

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinding by randomization schedule
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo + IV Meropenem (Placebo Comparator): Placebo, oral administration, 4 times per day (q6h), beginning on day +1 after HCT until 72-hours after completion of IV Meropenem (MER)
  Interventions: Biological: SYN-004, Ribaxamase or Placebo
- SYN-004 + IV Meropenem (Active Comparator): SYN-004, oral administration, 150mg, 4 times per day (q6h), beginning on day +1 after HCT until 72-hours after completion of IV Meropenem (MER)
  Interventions: Biological: SYN-004, Ribaxamase or Placebo
- Placebo + IV Piperacillin/Tazobactam (Placebo Comparator): Placebo, oral administration, 4 times per day (q6h), beginning on day +1 after HCT until 72-hours after completion of IV Piperacillin/Tazobactam (PIP/TAZO)
  Interventions: Biological: SYN-004, Ribaxamase or Placebo
- SYN-004 + IV Piperacillin/Tazobactam (Active Comparator): SYN-004, oral administration, 150mg, 4 times per day (q6h), beginning on day +1 after HCT until 72-hours after completion of IV Piperacillin/Tazobactam (PIP/TAZO)
  Interventions: Biological: SYN-004, Ribaxamase or Placebo
- Placebo + IV Cefepime (Placebo Comparator): Placebo, oral administration, 4 times per day (q6h), beginning on day +1 after HCT until 72-hours after completion of IV Cefepime (FEP)
  Interventions: Biological: SYN-004, Ribaxamase or Placebo
- SYN-004 + Cefepime (Active Comparator): SYN-004, oral administration, 150mg, 4 times per day (q6h), beginning on day +1 after HCT until 72-hours after completion of IV Cefepime (FEP)
  Interventions: Biological: SYN-004, Ribaxamase or Placebo

INTERVENTIONS:
Biological: SYN-004, Ribaxamase or Placebo — SYN-004 is an oral formulation of a recombinant class-A beta-lactamase that hydrolyzes the beta-lactam ring of susceptible antibiotics that are excreted into the intestines

SUMMARY:
Study Objectives:

1. To evaluate the safety and tolerability of oral SYN-004 in adult allogeneic HCT (allo-HCT) recipients who develop fever after conditioning therapy and are treated with IV β-lactam antibiotics meropenem (MER), piperacillin tazobactam (PIP/TAZO), or cefepime (FEP).
2. To evaluate potential absorption of oral SYN-004 into the systemic circulation of allo-HCT recipients and potential SYN-004-mediated alterations to systemic levels and efficacy of IV MER, PIP/TAZO or FEP.
3. To evaluate potential protective effects of SYN-004 on the intestinal microbiome of allo-HCT recipients treated with IV MER, PIP/TAZO or FEP.
4. To obtain preliminary information on potential therapeutic benefits and patient outcomes of SYN-004 in allo-HCT recipients treated with IV MER, PIP/TAZO or FEP

DETAILED DESCRIPTION:
Study Design:

This is a single-center, placebo controlled, double blinded Phase 1b/2a study to assess the safety, tolerability and potential efficacy of orally administered SYN-004 in adult allo-HCT recipients. Participants will be randomized 2:1 to SYN-004 or placebo in blocks of three, stratified in three cohorts based on study assigned antibiotic (MER, piperacillin/tazobactam [PIP/TAZO], FEP) to be administered if the treating clinicians determine initiation of broad-spectrum antibiotics is indicated. As such, there will be six groups based on antibiotic cohort and randomized assignment of study drug:

Group 1: Placebo + IV MER (n=4) (MER control). Group 2: SYN-004 + IV MER (n=8) (MER treatment). Group 3: Placebo + IV PIP/TAZO (n=4) (PIP/TAZO control). Group 4: SYN-004 + IV PIP/TAZO (n=8) (PIP/TAZO treatment). Group 5: Placebo + IV FEP (n=4) (FEP control). Group 6: SYN-004 + IV FEP (n=8) (FEP treatment). Study-assigned antibiotics will be dosed as follows (adjusted for renal function as needed): MER 1 gram every 8 hours, PIP/TAZO 4.5 grams every 6 hours, FEP 1 gram every 8 hours. SYN-004 treated participants (Groups 2, 4 and 6) will be compared to control participants who receive placebo (Groups 1, 3 and 5, respectively). The study will be conducted in stages, commencing with Groups 1 and 2 who will be assigned to receive MER if antibiotics are indicated. MER is the first cohort because anti-infective efficacy of MER is not anticipated to be affected if SYN-004 is absorbed systemically. Accrual for Groups 3 and 4 (PIP/TAZO cohort) will begin only after review of the data from Groups 1 and 2 by the Data and Safety Monitoring Committee (DSMC) and agreement to proceed. PIP/TAZO is the next cohort because TAZO is a beta-lactamase inhibitor. As such, in the unlikely event of SYN-004 systemic absorption, TAZO systemic concentrations should be sufficient to inhibit any absorbed SYN-004. Accrual for the FEP cohort will begin after approval by the DSMC's review of results from groups 3 and 4.

Patients planned to receive an allo-HCT will be eligible for enrollment in the study and can be enrolled anytime from when it is known they will undergo HCT until day +1 after HCT (day of study drug start). Written informed consent will be obtained by all patients. To count towards the enrollment goal of 36 participants, a study participant must receive at least 80% of scheduled study drug doses from initiation of study assigned antibiotics through the second antibiotic pharmacokinetic assessment (7-9 days of concomitant study drug and study assigned antibiotic). Additional participants will be enrolled to replace participants who do not meet criteria to count towards the goal study enrollment until the goal enrollment is achieved.

This Phase 1b/2a study will use the SYN-004 dosing regimen (150 mg, PO, q6h) used in previous Phase 1 and Phase 2 clinical trials in healthy volunteers and patents with LRTIs. The first dose of study drug will be administered at day +1 after HCT and will be continued until Criteria for Discontinuation of Study Drug are met.

The study will consist of two periods: the Treatment Period and the Follow-up Period.

1. The Treatment Period will be defined as the time from first dose of study drug until the last dose. For participants who do not meet criteria for early discontinuation, study drug will be continued for 72 hours after last dose of MER, PIP/TAZO, or FEP.
2. The Follow-up Period begins after cessation of study drug dosing and is split into three parts:

   * Part A: up to 30 days after study drug was discontinued
   * Part B: from end of Part A to day +180 after HCT
   * Part C: from end of Part B to day +365 after HCT Patients enrolled in the study will receive conditioning and HCT according to their treatment plan. Fever and time of antibiotic start will be defined per local standard of care of patients. Cessation of antibiotic therapy and/or changes to antibiotic therapy will be at the discretion of the treating physician.

All participants will be evaluated as outlined in the Schedule of Assessments. At predetermined points during the study as outlined in the SOA, blood samples, urine samples, fecal swabs, and fecal samples will be collected for the indicated analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Participant provides written informed consent.
2. Male or female patients ≥18 years undergoing myeloablative allo-HCT for a hematologic malignancy or myeloproliferative disorder.
3. Participant is able to ingest the SYN-004 dosage form (size 0 hard capsule).

Exclusion Criteria:

1. Allergy(ies) to MER, PIP, TAZO, or FEP.
2. History of allergy to SYN-004 or its components.
3. Admitted for HCT and started on MER, PIP/TAZO, or FEP prior to enrollment in the present study.
4. Currently enrolled in another interventional clinical study or received an investigational drug or device within 30 days or within a time period consistent with a washout period of 5 half-lives before signing the Informed Consent Form, whichever is longer.
5. Recipients of umbilical cord blood transplantation.
6. Underlying condition requiring HCT is not in remission (per International Working Group definitions), except for myelodysplastic syndrome and lymphoma, as long as these conditions are chemotherapy responsive.
7. Creatinine clearance <60 mL/min/1.73 m² by Cockroft-Gault calculation.
8. Cardiac ejection fraction <50%.
9. Cirrhosis, bilirubin >1.5x upper limit of normal, or AST/ALT >2.5x upper limit of normal.
10. History of veno-occlusive disease (VOD) or hepatic sinusoidal obstructive syndrome (SOS).
11. DLCO and/or FEV1 ≤80% of normal.
12. Chronic HIV or HBV infection.
13. Invasive fungal infection not responding to treatment at time of HCT.
14. Known active bacterial or viral infection at time of HCT.
15. CDI in the preceding 6 months.
16. Unable to comply with study protocol as determined by primary investigator.
17. Active gastrointestinal (GI) bleeding at time of HCT.
18. Prior colectomy or short gut syndrome.
19. Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
SYN-004 systemic absorption | No more than 28 days
  Assess potential SYN-004 systemic absorption (if any) by measuring SYN-004 plasma concentrations
Systemic antibiotic concentrations | Up to 8 hours after IV administration of antibiotic
  Assess potential effects of SYN-004 on systemic antibiotic concentrations by measuring MER, PIP and FEP plasma levels and determining the area under the curve for antibiotic concentrations and time (T) of antibiotic concentration above the minimum inhibitory concentration (MIC) (T>MIC) using the Clinical and Laboratory Standards Institute (CLSI) MIC susceptibility breakpoint for Enterobacteriaceae and Pseudomonas aeruginosa for each individual participant
Bacteremia | Daily during treatment, and weekly until 30 days after discontinuation of SYN-004 or Placebo
  Assess the incidence of blood stream infections (bacteremia) with an organism susceptible to MER, PIP/TAZO or FEP while receiving SYN-004 concurrent with the antibiotic the organism is susceptible to, wherein the bacteremia is attributable to a clinical infection with adequate source control (if applicable) and unrelated to a device
Bacterial intestinal infections | Daily during treatment, and weekly until 30 days after discontinuation of SYN-004 or Placebo
  Assess the incidence and severity of bacterial intestinal infections other than CDI (such as typhlitis, neutropenic enterocolitis or diverticulitis) while on study drug and study assigned antibiotic
Grade 3 or 4 adverse events | Up to 30 days after the last dose of SYN-004 or Placebo
  Assess tolerability of SYN-004 and grade 3 or 4 adverse events up to 30 days after the last dose of SYN-004
Overall survival | Up to 30 days after the last dose of SYN-004 or Placebo
  Overall survival at 30 days after last dose of SYN-004

SECONDARY OUTCOMES:
First line failure of PIP/TAZO or FEP | Up to 30 days after the last dose of SYN-004 or Placebo
  Assess the number of study participants who fail first line PIP/TAZO or FEP therapy and require second line therapy with another antibiotic
Gut microbiome protection | Up to 30 days after the last dose of SYN-004 or Placebo, and up to 180 days after HCT
  Assess the ability of SYN-004 to protect the gut microbiome (defined by alterations from baseline in bacterial community composition, metabolic potential of the microbiome, and antibiotic resistome) in study participants treated with PIP/TAZO or FEP, and confirm lack of protection in study participants treated with MER at up to 30 days after last dose of SYN-004 (and up to 180 days after HCT)
Urine concentrations of 3-indoxyl sulfate | Up to 30 days after the last dose of SYN-004 or Placebo, and up to 180 days after HCT
  Assess urine concentrations of 3-indoxyl sulfate as a biomarker of fecal levels of Clostridium and Enterococcus species up to 30 days after last dose of SYN-004 (and 180 days after HCT)
Impact on immunosuppressant dosing | Up to 30 days after the last dose of SYN-004 or Placebo, and up to 180 days after HCT
  Assess impact of SYN-004 on immunosuppressant dosing and levels obtained through routine care up to 30 days after last dose of SYN-004 (and 180 days after HCT)

OTHER OUTCOMES:
Long-term overall survival | 180 and 365 days after HCT
  Overall survival at 180 and 365 days after HCT
Relapse free survival | 180 and 365 days after HCT
  Relapse free survival at 30 days after last dose of SYN-004 (and 180 and 365 days after HCT)
Incidence of aGVHD | 30 days after last dose of SYN-004 or Placebo, and 180 days after HCT
  Incidence of aGVHD at 30 days after last dose of SYN-004 (and 180 days after HCT)
GVHD and relapse free survival | 30 days after last dose of SYN-004 or Placebo, and 180 and 365 days after HCT
  GVHD and relapse free survival at 30 days after last dose of SYN-004 (and 180 and 365 days after HCT)
Incidence of CDI | 30 days after last dose of SYN-004 or Placebo, and up to 180 days after HCT
  Assess the incidence of CDI up to 30 days after last dose of SYN-004 (and up to 180 days after HCT)
Incidence of MDRO bacteremia and Candidemia | 30 days after last dose of SYN-004 or Placebo, and up to 180 days after HCT
  Assess the incidence of MDRO bacteremia and Candidemia up to 30 days after last dose of SYN-004 (and up to 180 days after HCT)
Incidence of chronic GVHD | 180 days and 1 year after HCT
  Assess incidence of chronic GVHD at 180 days and 1 year after HCT
New stool colonization with MDRO and Candida species | Up to 30 days after last dose of SYN-004 or Placebo, and up to 180 days after HCT
  Assess the rate of new stool colonization with MDRO and Candida species up to 30 days after last dose of SYN-004 (and up to 180 days after HCT)
Microbiome domination due to MDRO | Up to 30 days after last dose of SYN-004 or Placebo, and up to 180 days after HCT
  Assess microbiome domination (defined as ≥30% of all bacterial species present in the intestinal microbiome) due to MDRO up to 30 days after last dose of SYN-004 (and 180 days after HCT)
New colonization with C. difficile | Up to 30 days after last dose of SYN-004 or Placebo, and up to 180 days after HCT
  Assess new colonization with C. difficile

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No